CLINICAL TRIAL: NCT03139344
Title: Long Duration Activity and Metabolic Control After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard K Shields (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Richard K Shields, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 201503732; R01HD082109 (NIH)
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-01

CONDITIONS: Spinal Cord Injuries
Keywords: metabolism; exercise; glucose; secondary health conditions; quality of life
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Acute gene regulation: low frequency (Experimental): Adaptations in gene regulation in response to single-session low-frequency exercise.
  Interventions: Other: Low-frequency Exercise
- Acute gene regulation: high frequency (Experimental): Adaptations in gene regulation in response to single-session high-frequency exercise.
  Interventions: Other: High-frequency Exercise
- Training study: low frequency (Experimental): Adaptations in gene regulation, systemic metabolic markers, and patient-report metrics in response to training with low-frequency exercise.
  Interventions: Other: Low-frequency Exercise
- Training study: high frequency (Experimental): Adaptations in gene regulation in response to training with high-frequency exercise.
  Interventions: Other: High-frequency Exercise
- Comparator cohort (No Intervention): Participants will undergo selected outcome measures to provide comparison values for Experimental arms.

INTERVENTIONS:
Other: Low-frequency Exercise — The quadriceps/hamstrings will perform exercise via the application of low-frequency electrical stimulation.
  Arms: Acute gene regulation: low frequency; Training study: low frequency
Other: High-frequency Exercise — The quadriceps/hamstrings will perform exercise via the application of high-frequency electrical stimulation.
  Arms: Acute gene regulation: high frequency; Training study: high frequency

SUMMARY:
Skeletal muscle is the largest endocrine organ in the body, playing an indispensable role in glucose homeostasis. Spinal cord injury (SCI) prevents skeletal muscle from carrying out this important function. Dysregulation of glucose metabolism precipitates high rates of metabolic syndrome, diabetes, and other secondary health conditions (SHCs) of SCI. These SHCs exert a negative influence on health-related quality of life (HRQOL). New discoveries support that a low level of activity throughout the day offers a more effective metabolic stimulus than brief, episodic exercise bouts. The proposed study will translate this emerging concept to the population of individuals with SCI by using low-force, long-duration electrical muscle stimulation to subsidize daily activity levels. Recently, we demonstrated that this type of stimulation up-regulates key genes that foster an oxidative, insulin-sensitive phenotype in paralyzed muscle. We will now test whether this type of activity can improve glucose homeostasis and metabolic function in patients with chronic paralysis. We hypothesize that improvements in metabolic function will be accompanied by a reduction in SHCs and a concomitant improvement in self-reported HRQOL. The long-term goal of this research is to develop a rehabilitation strategy to protect the musculoskeletal health, metabolic function, and health-related quality of life of people living with complete SCI.

DETAILED DESCRIPTION:
Skeletal muscle is a critical organ for regulating glucose and insulin in the body as a whole, and post-spinal cord injury (SCI) adaptations in muscle severely undermine this capacity. Contemporary SCI rehabilitation for people with complete SCI does not intervene to protect the function of paralyzed skeletal muscle as a key regulator of metabolic homeostasis. Through its deleterious effects on multiple systems, metabolic disease is one of the leading sources of morbidity, mortality, and health care cost for this population.

In the non-SCI population, pervasive, frequent, low-magnitude muscle contractions can increase energy expenditure by 50.3% above sitting levels. The loss of this component of muscle activity contributes to the energy imbalance and metabolic dysregulation observed in SCI. Subsidizing low-magnitude muscle contractions may offer an important metabolic stimulus for people with SCI. The significance of this study is that it builds on previous work demonstrating healthful transcriptional and translational gene adaptations in response to electrical stimulation training in SCI. These adaptations may initiate improvements in systemic biomarkers of metabolic health and improvements in secondary health conditions and health-related quality of life.

In our previous work, we demonstrated that regular electrical stimulation of paralyzed muscle up-regulates PGC-1α, a key transcriptional co-activator for skeletal muscle and metabolic adaptation. Our previous work also indicates that electrical stimulation alters the expression of genes controlling mitochondrial biogenesis. However, we understand very little about the optimal amount of electrically-evoked muscle activity to deliver in order to promote positive metabolic adaptations. Long duration, low force contractions are likely to be most advantageous for promoting metabolic stability in people with chronic SCI, who also have osteoporosis and are unable to receive high force muscle contractions induced by conventional rehabilitation protocols. This study will intervene with a protocol of low-force, long-duration muscle stimulation designed to instigate systemic metabolic adaptations. In the proposed study we hypothesize that gene-level adaptations will yield tissue-level improvements in glucose utilization that facilitate systemic improvements in clinical markers of metabolic control, culminating in fewer secondary health conditions and enhanced health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Motor complete SCI (AIS A-B)

Exclusion Criteria:

* Pressure ulcers, chronic infection, lower extremity muscle contractures, deep vein thrombosis, bleeding disorder, recent limb fractures, pregnancy, metformin or other medications for diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Shields, PhD, PT, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dudley-Javoroski S, Saha PK, Liang G, Li C, Gao Z, Shields RK. High dose compressive loads attenuate bone mineral loss in humans with spinal cord injury. Osteoporos Int. 2012 Sep;23(9):2335-46. doi: 10.1007/s00198-011-1879-4. Epub 2011 Dec 21. PMID 22187008
- [Background] Dudley-Javoroski S, Shields RK. Dose estimation and surveillance of mechanical loading interventions for bone loss after spinal cord injury. Phys Ther. 2008 Mar;88(3):387-96. doi: 10.2522/ptj.20070224. Epub 2008 Jan 17. PMID 18202080
- [Background] Dudley-Javoroski S, Shields RK. Active-resisted stance modulates regional bone mineral density in humans with spinal cord injury. J Spinal Cord Med. 2013 May;36(3):191-9. doi: 10.1179/2045772313Y.0000000092. PMID 23809588
- [Background] Dudley-Javoroski S, Littmann AE, Iguchi M, Shields RK. Doublet stimulation protocol to minimize musculoskeletal stress during paralyzed quadriceps muscle testing. J Appl Physiol (1985). 2008 Jun;104(6):1574-82. doi: 10.1152/japplphysiol.00892.2007. Epub 2008 Apr 24. PMID 18436697
- [Background] Dudley-Javoroski S, Shields RK. Assessment of physical function and secondary complications after complete spinal cord injury. Disabil Rehabil. 2006 Jan 30;28(2):103-10. doi: 10.1080/09638280500163828. PMID 16393840
- [Background] Adams CM, Suneja M, Dudley-Javoroski S, Shields RK. Altered mRNA expression after long-term soleus electrical stimulation training in humans with paralysis. Muscle Nerve. 2011 Jan;43(1):65-75. doi: 10.1002/mus.21831. PMID 21171097
- [Background] Frey Law LA, Shields RK. Femoral loads during passive, active, and active-resistive stance after spinal cord injury: a mathematical model. Clin Biomech (Bristol). 2004 Mar;19(3):313-21. doi: 10.1016/j.clinbiomech.2003.12.005. PMID 15003348
- [Background] Kunkel SD, Suneja M, Ebert SM, Bongers KS, Fox DK, Malmberg SE, Alipour F, Shields RK, Adams CM. mRNA expression signatures of human skeletal muscle atrophy identify a natural compound that increases muscle mass. Cell Metab. 2011 Jun 8;13(6):627-38. doi: 10.1016/j.cmet.2011.03.020. PMID 21641545
- [Background] McHenry CL, Wu J, Shields RK. Potential regenerative rehabilitation technology: implications of mechanical stimuli to tissue health. BMC Res Notes. 2014 Jun 3;7:334. doi: 10.1186/1756-0500-7-334. PMID 24894666
- [Background] McHenry CL, Shields RK. A biomechanical analysis of exercise in standing, supine, and seated positions: Implications for individuals with spinal cord injury. J Spinal Cord Med. 2012 May;35(3):140-7. doi: 10.1179/2045772312Y.0000000011. PMID 22507023
- [Background] Petrie MA, Suneja M, Faidley E, Shields RK. A minimal dose of electrically induced muscle activity regulates distinct gene signaling pathways in humans with spinal cord injury. PLoS One. 2014 Dec 22;9(12):e115791. doi: 10.1371/journal.pone.0115791. eCollection 2014. PMID 25531450
- [Background] Petrie MA, Suneja M, Faidley E, Shields RK. Low force contractions induce fatigue consistent with muscle mRNA expression in people with spinal cord injury. Physiol Rep. 2014 Feb 25;2(2):e00248. doi: 10.1002/phy2.248. eCollection 2014 Feb 1. PMID 24744911
- [Background] Shields RK, Dudley-Javoroski S. Monitoring standing wheelchair use after spinal cord injury: a case report. Disabil Rehabil. 2005 Feb 4;27(3):142-6. doi: 10.1080/09638280400009337. PMID 15823996
- [Background] Petrie M, Suneja M, Shields RK. Low-frequency stimulation regulates metabolic gene expression in paralyzed muscle. J Appl Physiol (1985). 2015 Mar 15;118(6):723-31. doi: 10.1152/japplphysiol.00628.2014. Epub 2015 Jan 29. PMID 25635001
- [Background] Zhorne R, Dudley-Javoroski S, Shields RK. Skeletal muscle activity and CNS neuro-plasticity. Neural Regen Res. 2016 Jan;11(1):69-70. doi: 10.4103/1673-5374.169623. No abstract available. PMID 26981083
- [Background] Petrie MA, Kimball AL, McHenry CL, Suneja M, Yen CL, Sharma A, Shields RK. Distinct Skeletal Muscle Gene Regulation from Active Contraction, Passive Vibration, and Whole Body Heat Stress in Humans. PLoS One. 2016 Aug 3;11(8):e0160594. doi: 10.1371/journal.pone.0160594. eCollection 2016. PMID 27486743
- [Background] Shields RK. Turning Over the Hourglass. Phys Ther. 2017 Oct 1;97(10):949-963. doi: 10.1093/ptj/pzx072. PMID 29029555
- [Background] Woelfel JR, Kimball AL, Yen CL, Shields RK. Low-Force Muscle Activity Regulates Energy Expenditure after Spinal Cord Injury. Med Sci Sports Exerc. 2017 May;49(5):870-878. doi: 10.1249/MSS.0000000000001187. PMID 28009786
- [Background] Yen CL, McHenry CL, Petrie MA, Dudley-Javoroski S, Shields RK. Vibration training after chronic spinal cord injury: Evidence for persistent segmental plasticity. Neurosci Lett. 2017 Apr 24;647:129-132. doi: 10.1016/j.neulet.2017.03.019. Epub 2017 Mar 16. PMID 28315725
- [Background] Oza PD, Dudley-Javoroski S, Shields RK. Modulation of H-Reflex Depression with Paired-Pulse Stimulation in Healthy Active Humans. Rehabil Res Pract. 2017;2017:5107097. doi: 10.1155/2017/5107097. Epub 2017 Oct 31. PMID 29225972
- [Background] Woelfel JR, Dudley-Javoroski S, Shields RK. Precision Physical Therapy: Exercise, the Epigenome, and the Heritability of Environmentally Modified Traits. Phys Ther. 2018 Nov 1;98(11):946-952. doi: 10.1093/ptj/pzy092. PMID 30388254
- [Background] Cole KR, Dudley-Javoroski S, Shields RK. Hybrid stimulation enhances torque as a function of muscle fusion in human paralyzed and non-paralyzed skeletal muscle. J Spinal Cord Med. 2019 Sep;42(5):562-570. doi: 10.1080/10790268.2018.1485312. Epub 2018 Jun 20. PMID 29923814
- [Background] Dudley-Javoroski S, Lee J, Shields RK. Cognitive function, quality of life, and aging: relationships in individuals with and without spinal cord injury. Physiother Theory Pract. 2022 Jan;38(1):36-45. doi: 10.1080/09593985.2020.1712755. Epub 2020 Jan 8. PMID 31914347
- [Background] Petrie MA, Sharma A, Taylor EB, Suneja M, Shields RK. Impact of short- and long-term electrically induced muscle exercise on gene signaling pathways, gene expression, and PGC1a methylation in men with spinal cord injury. Physiol Genomics. 2020 Feb 1;52(2):71-80. doi: 10.1152/physiolgenomics.00064.2019. Epub 2019 Dec 23. PMID 31869286
- [Background] Lee J, Dudley-Javoroski S, Shields RK. Motor demands of cognitive testing may artificially reduce executive function scores in individuals with spinal cord injury. J Spinal Cord Med. 2021 Mar;44(2):253-261. doi: 10.1080/10790268.2019.1597482. Epub 2019 Apr 3. PMID 30943119
- [Background] Shields RK. Precision Rehabilitation: How Lifelong Healthy Behaviors Modulate Biology, Determine Health, and Affect Populations. Phys Ther. 2022 Jan 1;102(1):pzab248. doi: 10.1093/ptj/pzab248. No abstract available. PMID 34718793
- [Background] Shields RK, Dudley-Javoroski S. Epigenetics and the International Classification of Functioning, Disability and Health Model: Bridging Nature, Nurture, and Patient-Centered Population Health. Phys Ther. 2022 Jan 1;102(1):pzab247. doi: 10.1093/ptj/pzab247. PMID 34718813
- [Background] Petrie MA, Taylor EB, Suneja M, Shields RK. Genomic and Epigenomic Evaluation of Electrically Induced Exercise in People With Spinal Cord Injury: Application to Precision Rehabilitation. Phys Ther. 2022 Jan 1;102(1):pzab243. doi: 10.1093/ptj/pzab243. PMID 34718779

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acute Gene Regulation: Low Frequency | Acute Gene Regulation: High Frequency | Training Study: Low Frequency | Training Study: High Frequency | Comparator Cohort
Started | 28 | 12 | 21 | 10 | 18
Completed | 28 | 12 | 21 | 10 | 18
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acute Gene Regulation: Low Frequency | Acute Gene Regulation: High Frequency | Training Study: Low Frequency | Training Study: High Frequency | Comparator Cohort | Total
Number analyzed (Participants) | 28 | 12 | 21 | 10 | 18 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 12 | 21 | 10 | 18 | 89
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 8 | 3 | 4 | 29
  Male | 18 | 8 | 13 | 7 | 14 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 27 | 12 | 21 | 10 | 17 | 87
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 2 | 0 | 2 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 0 | 1 | 5
  White | 23 | 11 | 18 | 10 | 17 | 79
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 12 | 21 | 10 | 18 | 89
Quadriplegia versus Paraplegia [Count of Participants; unit: Participants]
  Quadriplegia | 8 | 4 | 6 | 2 | 6 | 26
  Paraplegia | 20 | 8 | 15 | 8 | 12 | 63

OUTCOME MEASURES:

1. Primary Outcome: Acute Gene Regulation: NR4A3 mRNA Expression Pre and Post-Stimulation
Description: Acute post-stimulation effect upon skeletal muscle nuclear receptor subfamily 4 group A member 3 (NR4A3) expression, measured via muscle biopsy and exon array analysis. Probe summarization and probe set normalization were performed using robust multichip average, which included background correction, quantile normalization, log2 transformation and median polish probe set summarization. 0 represents no mRNA expression and higher values represent greater expression compared to all genes in the microarray.
Time Frame: 3 hours after a single session of electrical stimulation
Population: This outcome measure only pertains to the single-session (3 hour) study arms: Acute Gene Regulation: Low Frequency and Acute Gene Regulation: High Frequency
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Acute Gene Regulation: Low Frequency | Acute Gene Regulation: High Frequency
Number analyzed (Participants) | 28 | 12
arbitrary units
  Pre-Stimulation | 3.235 (0.81) | 2.711 (0.49)
  Post-Stimulation | 6.286 (0.78) | 5.772 (0.49)
Statistical Analysis 1: Comparison: Acute Gene Regulation: Low Frequency; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Acute Gene Regulation: High Frequency; Test type: Superiority; p < 0.001, ANOVA

2. Primary Outcome: Acute Gene Regulation: PGC1-alpha mRNA Expression Pre and Post-Stimulation
Description: Acute post-stimulation effect upon skeletal muscle peroxisome proliferator-activated gamma coactivator (PGC1-alpha) expression, measured via muscle biopsy and exon array analysis. Probe summarization and probe set normalization were performed using robust multichip average, which included background correction, quantile normalization, log2 transformation and median polish probe set summarization. 0 represents no mRNA expression and higher values represent greater expression compared to all genes in the microarray.
Time Frame: 3 hours after a single session of electrical stimulation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Acute Gene Regulation: Low Frequency | Acute Gene Regulation: High Frequency
Number analyzed (Participants) | 28 | 12
arbitrary units
  Pre-Stimulation | 5.37 (0.48) | 4.92 (0.30)
  Post-Stimulation | 6.72 (0.39) | 6.43 (0.30)
Statistical Analysis 1: Comparison: Acute Gene Regulation: Low Frequency; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Acute Gene Regulation: High Frequency; Test type: Superiority; p < 0.001, ANOVA

3. Primary Outcome: Acute Gene Regulation: ABRA mRNA Expression Pre and Post-Stimulation
Description: Acute post-stimulation effect upon skeletal muscle actin binding Rho activating protein (ABRA) expression, measured via muscle biopsy and exon array analysis. Probe summarization and probe set normalization were performed using robust multichip average, which included background correction, quantile normalization, log2 transformation and median polish probe set summarization. 0 represents no mRNA expression and higher values represent greater expression compared to all genes in the microarray.
Time Frame: 3 hours after a single session of electrical stimulation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Acute Gene Regulation: Low Frequency | Acute Gene Regulation: High Frequency
Number analyzed (Participants) | 28 | 12
arbitrary units
  Pre-Stimulation | 6.76 (0.993) | 5.63 (0.34)
  Post-Stimulation | 8.61 (0.76) | 7.71 (0.34)
Statistical Analysis 1: Comparison: Acute Gene Regulation: Low Frequency; Test type: Superiority; p = 0.011, ANOVA
Statistical Analysis 2: Comparison: Acute Gene Regulation: High Frequency; Test type: Superiority; p < 0.001, ANOVA

4. Primary Outcome: Acute Gene Regulation: PDK4 mRNA Expression Pre and Post-Stimulation
Description: Acute post-stimulation effect upon skeletal muscle pyruvate dehydrogenase kinase 4 (PDK4) expression, measured via muscle biopsy and exon array analysis. Probe summarization and probe set normalization were performed using robust multichip average, which included background correction, quantile normalization, log2 transformation and median polish probe set summarization. 0 represents no mRNA expression and higher values represent greater expression compared to all genes in the microarray.
Time Frame: 3 hours after a single session of electrical stimulation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Acute Gene Regulation: Low Frequency | Acute Gene Regulation: High Frequency
Number analyzed (Participants) | 28 | 12
arbitrary units
  Pre-Stimulation | 6.64 (0.38) | 6.46 (0.44)
  Post-Stimulation | 7.23 (0.38) | 7.45 (0.44)
Statistical Analysis 1: Comparison: Acute Gene Regulation: Low Frequency; Test type: Superiority; p = 0.148, ANOVA
Statistical Analysis 2: Comparison: Acute Gene Regulation: High Frequency; Test type: Superiority; p = 0.005, ANOVA

5. Primary Outcome: Post-training Gene Regulation: MYH6 mRNA Expression Baseline and Post-Training
Description: Pre- and post-training skeletal muscle myosin heavy chain 6 (MYH6) expression, measured via muscle biopsy and exon array analysis. Probe summarization and probe set normalization were performed using robust multichip average, which included background correction, quantile normalization, log2 transformation and median polish probe set summarization. 0 represents no mRNA expression and higher values represent greater expression compared to all genes in the microarray.
Time Frame: 6 months
Population: This outcome measure only pertains to the Training study arms: Training Study: Low Frequency and Training Study: High Frequency.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Training Study: Low Frequency | Training Study: High Frequency
Number analyzed (Participants) | 21 | 10
arbitrary units
  Baseline | 6.61 (0.71) | 5.38 (0.69)
  Post-Training | 7.10 (0.88) | 6.58 (0.69)
Statistical Analysis 1: Comparison: Training Study: Low Frequency; Test type: Superiority; p = 0.069, ANOVA
Statistical Analysis 2: Comparison: Training Study: High Frequency; Test type: Superiority; p = 0.003, ANOVA

6. Primary Outcome: Post-training Gene Regulation: MYL3 mRNA Expression Baseline and Post-Training
Description: Pre- and post-training skeletal muscle myosin light chain 3 (MYL3) expression, measured via muscle biopsy and exon array analysis. Probe summarization and probe set normalization were performed using robust multichip average, which included background correction, quantile normalization, log2 transformation and median polish probe set summarization. 0 represents no mRNA expression and higher values represent greater expression compared to all genes in the microarray.
Time Frame: 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Training Study: Low Frequency | Training Study: High Frequency
Number analyzed (Participants) | 21 | 10
arbitrary units
  Baseline | 7.37 (0.87) | 6.38 (0.81)
  Post-Training | 8.01 (1.08) | 7.96 (0.81)
Statistical Analysis 1: Comparison: Training Study: Low Frequency; Test type: Superiority; p = 0.118, ANOVA
Statistical Analysis 2: Comparison: Training Study: High Frequency; Test type: Superiority; p = 0.010, ANOVA

7. Primary Outcome: Post-training Gene Regulation: MYH7 mRNA Expression Baseline and Post-Training
Description: Pre- and post-training skeletal muscle myosin heavy chain 7 (MYH7) expression, measured via muscle biopsy and exon array analysis. Probe summarization and probe set normalization were performed using robust multichip average, which included background correction, quantile normalization, log2 transformation and median polish probe set summarization. 0 represents no mRNA expression and higher values represent greater expression compared to all genes in the microarray.
Time Frame: 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Training Study: Low Frequency | Training Study: High Frequency
Number analyzed (Participants) | 21 | 10
arbitrary units
  Baseline | 8.55 (1.1) | 7.16 (0.88)
  Post-Training | 9.43 (1.4) | 8.85 (0.88)
Statistical Analysis 1: Comparison: Training Study: Low Frequency; Test type: Superiority; p = 0.059, ANOVA
Statistical Analysis 2: Comparison: Training Study: High Frequency; Test type: Superiority; p = 0.015, ANOVA

8. Primary Outcome: Post-training Gene Regulation: ACTN3 mRNA Expression Baseline and Post-Training
Description: Pre- and post-training skeletal muscle actin 3 (ACTN3) expression, measured via muscle biopsy and exon array analysis. Probe summarization and probe set normalization were performed using robust multichip average, which included background correction, quantile normalization, log2 transformation and median polish probe set summarization. 0 represents no mRNA expression and higher values represent greater expression compared to all genes in the microarray.
Time Frame: 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Training Study: Low Frequency | Training Study: High Frequency
Number analyzed (Participants) | 21 | 10
arbitrary units
  Baseline | 8.95 (0.79) | 8.51 (0.74)
  Post-Training | 8.20 (0.71) | 7.12 (0.74)
Statistical Analysis 1: Comparison: Training Study: Low Frequency; Test type: Superiority; p = 0.010, ANOVA
Statistical Analysis 2: Comparison: Training Study: High Frequency; Test type: Superiority; p = 0.001, ANOVA

9. Primary Outcome: Post-training Metabolism: Fasting Insulin
Description: Pre- and post-training fasting insulin, measured via venipuncture and standard laboratory assays
Time Frame: 6 months
Population: This outcome measure only pertains to the Training Study: Low Frequency arm. 11 participants contributed venous blood samples.
Measure: Mean (Standard Deviation); unit: microU/mL
Arm/Group | Training Study: Low Frequency
Number analyzed (Participants) | 11
microU/mL
  Pre-Training | 19.245 (16.387)
  Post-Training | 8.305 (3.407)
Statistical Analysis 1: Comparison: Training Study: Low Frequency; Test type: Superiority; p = 0.036, t-test, 2 sided

10. Primary Outcome: Post-training Metabolism: Fasting Glucose
Description: Pre- and post-training fasting glucose, measured via venipuncture and standard laboratory assays
Time Frame: 6 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Training Study: Low Frequency
Number analyzed (Participants) | 11
mg/dL
  Pre-Training | 94.727 (10.725)
  Post-Training | 91.091 (14.223)
Statistical Analysis 1: Comparison: Training Study: Low Frequency; Test type: Superiority; p = 0.345, t-test, 2 sided

11. Primary Outcome: Post-training Metabolism: Fasting Glucose-insulin Ratio
Description: Pre- and post-training ratio of fasting glucose to fasting insulin, measured via venipuncture and standard laboratory assays
Time Frame: 6 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Training Study: Low Frequency
Number analyzed (Participants) | 11
ratio
  Pre-Training | 8.649 (5.573)
  Post-Training | 11.274 (5.417)
Statistical Analysis 1: Comparison: Training Study: Low Frequency; Test type: Superiority; p = 0.264, t-test, 2 sided

12. Primary Outcome: Post-training Metabolism: Fasting Hemoglobin A1c (HBA1c)
Description: Pre- and post-training fasting Hemoglobin A1C (HbA1c), measured via venipuncture and standard laboratory assays
Time Frame: 6 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent of total hemoglobin
Arm/Group | Training Study: Low Frequency
Number analyzed (Participants) | 11
percent of total hemoglobin
  Pre-training | 4.227 (1.030)
  Post-training | 3.970 (0.946)
Statistical Analysis 1: Comparison: Training Study: Low Frequency; Test type: Superiority; p = 0.266, t-test, 2 sided

13. Primary Outcome: Post-training Metabolism: C-reactive Protein (CRP)
Description: Pre- and post-training C-reactive protein (CRP), measured via venipuncture and standard laboratory assays
Time Frame: 6 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Training Study: Low Frequency
Number analyzed (Participants) | 11
mg/L
  Pre-training | 11.427 (11.137)
  Post-training | 4.545 (2.581)
Statistical Analysis 1: Comparison: Training Study: Low Frequency; Test type: Superiority; p = 0.040, t-test, 2 sided

14. Primary Outcome: Pre-training Subject-report Measures: PROMIS Physical Health
Description: Pre-training Patient Reported Outcomes Measurement Information Systems (PROMIS) Global Health - Physical health T-score
  Theoretical minimum = 16.2, Theoretical maximum = 67.7, higher scores signify more of the construct being measured (eg. physical health). US population mean = 50, SD = 10.
Time Frame: Baseline
Population: This outcome measure pertained only to the Training Study: Low Frequency arm and to the Comparator Cohort. 11 participants in the Training study: low frequency arm contributed PROMIS subject-report measures.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Training Study: Low Frequency | Comparator Cohort
Number analyzed (Participants) | 11 | 18
T-score | 39.9 (4.9) | 37.0 (4.1)
Statistical Analysis 1: Comparison: Training Study: Low Frequency vs Comparator Cohort; Test type: Superiority; p = 0.109, t-test, 2 sided

15. Primary Outcome: Pre-training Subject Report Measures: PROMIS Mental Health
Description: Pre-training Patient Reported Outcomes Measurement Information Systems (PROMIS) Global Health - Mental health T-score
  Theoretical minimum = 21.2, Theoretical maximum = 67.6, higher scores signify more of the construct being measured (eg. mental health). US population mean = 50, SD = 10.
Time Frame: Baseline
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Training Study: Low Frequency | Comparator Cohort
Number analyzed (Participants) | 11 | 18
T-score | 47.0 (5.1) | 47.3 (4.1)
Statistical Analysis 1: Comparison: Training Study: Low Frequency vs Comparator Cohort; Test type: Superiority; p = 0.895, t-test, 2 sided

16. Primary Outcome: Post-training Subject-report Measures: PROMIS Physical Health
Description: Pre- and post-training Patient Reported Outcomes Measurement Information Systems (PROMIS) Global Health - Physical health T-score
  Theoretical minimum = 16.2, Theoretical maximum = 67.7, higher scores signify more of the construct being measured (eg. physical health). US population mean = 50, SD = 10.
Time Frame: 6 months
Population: This outcome measure pertained only to the Training Study: Low Frequency arm. 11 participants contributed PROMIS subject-report measures.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Training Study: Low Frequency
Number analyzed (Participants) | 11
T-score
  Pre-training | 39.9 (4.9)
  Post-training | 39.5 (5.6)
Statistical Analysis 1: Comparison: Training Study: Low Frequency; Test type: Superiority; p = 0.573, t-test, 2 sided; paired t-test

17. Primary Outcome: Post-training Subject-report Measures: PROMIS Mental Health
Description: Pre- and post-training Patient Reported Outcomes Measurement Information Systems (PROMIS) Global Health - Mental health T-score
  Theoretical minimum = 21.2, Theoretical maximum = 67.6, higher scores signify more of the construct being measured (eg. mental health). US population mean = 50, SD = 10.
Time Frame: 6 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Training Study: Low Frequency
Number analyzed (Participants) | 11
T-score
  Pre-training | 47.0 (5.1)
  Post-training | 47.3 (5.1)
Statistical Analysis 1: Comparison: Training Study: Low Frequency; Test type: Superiority; p = 0.858, t-test, 2 sided; paired t-test

ADVERSE EVENTS:
Time Frame: From Baseline to 6 months
Arm/Group | Acute Gene Regulation: Low Frequency | Acute Gene Regulation: High Frequency | Training Study: Low Frequency | Training Study: High Frequency | Comparator Cohort
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/12 | 0/21 | 0/10 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/12 | 0/21 | 0/10 | 0/18
Other Adverse Events (participants affected / at risk) | 0/28 | 0/12 | 0/21 | 0/10 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT03139344/Prot_SAP_000.pdf